CLINICAL TRIAL: NCT05805982
Title: Randomized Non Inferiority Trial of Educational Video Versus In-person Genetic Counseling for Hereditary Cancer
Brief Title: Educational Video Versus In-person Genetic Counseling for Hereditary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Yanin Chavarri Guerra, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HEM-3442
Record Dates: First submitted 2023-02-07; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Genetic Counseling; Hereditary Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video (Experimental): The patient will watch a 15-minute video on an electronic tablet that includes the following items:
  * What is hereditary cancer?
  * Inheritance risk
  * Who are candidates for a genetic test?
  * What is a genetic testing and how can it help?
  * What types of results can be expected from genetic testing?
  * Reactions to the result of the genetic test
  * Clinical care according to the results
  * Any common questions? When the patient finish watching the video, he/she would have the opportunity to resolve any doubts.
  Interventions: Behavioral: Educational Video
- In-Person genetic counseling (Active Comparator): Patients will receive pre-test genetic counseling in person with a specialist using the usual protocols existing at the Institute and systematically includes the following:
  Family history of cancer Personal cancer risk assessment Education on inheritance and disease expression Types of tests and results (positive, negative and variants of uncertain significance).
  Limitations of the genetic study Preparation of possible outcomes according to results Risks Additional information: confidentiality of the results, costs and test options. Opportunity will be given to resolve doubts
  Interventions: Behavioral: In person genetic cancer counseling

INTERVENTIONS:
Behavioral: Educational Video — Pre-recorded educational video including hereditary cancer information, genetic cancer testing candidates, types of testing, type of results, benefits and risks, recommendations according to results, inheritance and common questions.
  Arms: Educational Video
Behavioral: In person genetic cancer counseling — Includes:
  Family history of cancer (3-generation family tree) Personal Cancer Risk Assessment Education on inheritance and expression of disease Types of tests Preparation on possible outcomes according to results Obtaining consent for test Opportunity to solve doubts
  Arms: In-Person genetic counseling

SUMMARY:
The identification of mutations in cancer susceptibility genes is important as it makes it possible to recommend specific cancer treatments, implement risk reduction strategies or early detection of cancer, and identify family members at risk. The guidelines for evaluating patients who are candidates for genetic testing recommend pre-test genetic counseling. However, the limited number of specialists trained to provide genetic counseling worldwide, and particularly in developing countries such as Mexico, makes it difficult to implement such recommendations. The present proposal aims to compare, through a randomized non-inferiority study, a pre-test education strategy using a pre-recorded video against in-person counseling. This strategy could potentially increase access in places with limited resources.

The general hypothesis of the research is that patients who are candidates for cancer genetic susceptibility testing who receive pre-test education via video will consent to genetic testing in the same proportion as those who receive it during an in-person visit.

The specific objectives of the study include: 1) to compare the proportion of patients who are tested in both groups; 2) to assess knowledge about hereditary cancer in both groups after the intervention; 3) assess anxiety symptoms in both groups after the intervention; and 4) assess satisfaction with the information received during the intervention.Patients >18 years of age who meet the criteria for genetic testing to evaluate genetic cancer susceptibility genes and who have not previously undergone genetic testing or genetic counseling will be invited. The intervention group will receive education via pre-recorded video and the control group will receive genetic counseling during an in-person consultation.

ELIGIBILITY:
Inclusion Criteria:

* Meet cancer genetic testing criteria

Exclusion Criteria:

* Had a genetic testing before
* Had genetic counseling before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Genetic testing acceptance | up to 12 weeks
  Proportion of patients that accept to undergo a genetic testing

SECONDARY OUTCOMES:
Genetic cancer knowledge change (pre and post intervention) | up to 24 hours after intervention
  Knowgene questionnaire
Anxiety level (pre and post intervention) | up to 24 hours after intervention
  GAD-7 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No